CLINICAL TRIAL: NCT00458419
Title: Role of Endorphins in the Perception of Dyspnea in Patients With Chronic Obstructive Pulmonary Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Diagnostic
Other Study IDs: 17355
Record Dates: First submitted 2007-04-08; First posted 2007-04-10 (Estimated); Last update posted 2007-11-02 (Estimated); Status verified 2007-10

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: dyspnea; leg discomfort; exercise duration
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Dyspnea | interventions — Naloxone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- A: naloxone; B: normal saline (Placebo Comparator): Arm A: IV naloxone Arm B: IV normal saline
  Interventions: Drug: naloxone versus placebo; Drug: intravenous injection of normal saline or naloxone

INTERVENTIONS:
Drug: naloxone versus placebo — 10 mg of naloxone administered IV or normal saline administered IV in randomized order at different visits
Drug: intravenous injection of normal saline or naloxone — Arm A: 10 mg of naloxone given IV in 25 ml of normal saline Arm B: 25 ml of normal saline

SUMMARY:
Endorphins are naturally occurring narcotic substances that are released when individuals perform exercise. The hypothesis of the study is that endorphins reduce the severity of breathlessness during exercise in patients with chronic obstructive pulmonary disease (COPD). The initial five visits include familiarization and validation of a computerized system for patients to report dyspnea and leg discomfort continuously during exercise testing.

At Visits 6 and 7 blood is drawn to measure serum endorphin levels pre-exercise, end exercise, and 30 minutes after exercise. Normal saline or naloxone is given intravenously 5 minutes prior to exercise in a double-blinded design. The primary outcome is the slope of oxygen consumption - dyspnea.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of COPD
* Ability to exercise
* Ability to computer mouse to provide ratings
* > 10 pack-years smoking
* Baseline dyspnea index < 9

Exclusion Criteria:

* Clinically significant comorbidities

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2005-09; Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Slope of oxygen consumption - dyspnea during treadmill exercise. | throughout exercise

SECONDARY OUTCOMES:
Exercise duration | 10-14 minutes
Peak ratings of breathlessness | at end of exercsie - 10-15 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Doanld A Mahler, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States

REFERENCES:
- [Derived] Mahler DA, Murray JA, Waterman LA, Ward J, Kraemer WJ, Zhang X, Baird JC. Endogenous opioids modify dyspnoea during treadmill exercise in patients with COPD. Eur Respir J. 2009 Apr;33(4):771-7. doi: 10.1183/09031936.00145208. Epub 2009 Feb 12. PMID 19213787